CLINICAL TRIAL: NCT05945758
Title: Esthetic and Clinical Assessment of Injectable Resin Composite Technique Compared to Conventional Layering Technique in Patients With Multiple Spacing in the Maxillary Anterior Teeth Area.
Brief Title: Esthetic and Clinical Assessment of Injectable Resin Composite Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tasneem Mokhtar Ali Morad, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Injection Molding Technique
Record Dates: First submitted 2023-07-04; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Clinical Performance
Keywords: injectable resin composite; conventional layering technique; FDI; multiple spacing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spacing in the maxillary anterior teeth area treated with injectable resin composite technique. (Experimental): The injectable composite resin technique is an indirect/direct method that uses a transparent silicone index for accurate and predictable translation of diagnostic wax-up into composite restorations without the need for tooth preparation.
  The Spaces will be restored with injectable resin composite.
  Interventions: Procedure: Injectable resin composite technique.
- Spacing in the maxillary anterior teeth area treated with conventional layering composite technique. (Active Comparator): shade mapping of enamel and dentin, then isolation the teeth with rubber dam. Palatal index will be done on waxing up and applied against the palatal surface to check the adaptation of the index. Then, the enamel shade adapted on the index in the spacing area. index will be placed back on the anterior teeth to build the palatal wall. A brush will be used to adapt the composite to the margin. After removing excess material, light curing will be carried out for 20 seconds. The Unica matrix (Polydentia) will be used to restore the proximal wall, and to achieve a good seal with the palatal wall. The matrix can be stabilized with a wedge if necessary. Building the proximal wall using the enamel shade, and the incisal halo by using a dentin shade, the frame to layer the core of the restoration will be ready.
  Interventions: Procedure: Conventional layering technique

INTERVENTIONS:
Procedure: Injectable resin composite technique. — A metal impression tray was filled with transparent vinyl polysiloxane (EXACLEAR, GC) and used to copy the stone model with the wax-up. Then, the replica will be separated from metal tray and a needle-shaped bur will be used to drill holes through the silicone key ending in the middle of the incisal edge. It will be checked whether the holes were large enough to enable the tip of the composite syringe to pass easily and completely. Neighbouring teeth (mesial and distal one) isolated using Teflon tape, as each tooth will individually be restored for establishment of satisfactory contact points. Following etching and rinsing, the tooth dried, and a dental cord (Ultrampak, Ultradent) will be packed into sulcus for mechanical prevention of subgingival composite flow. Then, the transparent silicone index will be placed in the correct intraoral position, and a syringe filled with flowable composite will be inserted through the hole on the incisal edge.
  Other Names: Beautiful Flow Plus F03, Medium Viscosity, Shofu Dental
  Arms: Spacing in the maxillary anterior teeth area treated with injectable resin composite technique.
Procedure: Conventional layering technique — the palatal surface will be restored by enamel shade; adapted on the index in the spacing area then The Unica matrix (Polydentia) will be used to restore the proximal wall, and to achieve a good seal with the palatal wall. The matrix can be stabilized with a wedge if necessary. Building the proximal wall using the enamel shade, and the incisal halo by using a dentin shade, the frame to layer the core of the restoration will be ready.
  Other Names: Enamel and Dentin shades
  Arms: Spacing in the maxillary anterior teeth area treated with conventional layering composite technique.

SUMMARY:
injectable resin composite technique will show a better clinical and esthetic performance compared to conventional layering resin composite technique in patients with multiple spacing in the maxillary anterior teeth area or not.

DETAILED DESCRIPTION:
The injectable composite resin technique is an indirect/direct method that uses a transparent silicone index for accurate and predictable translation of diagnostic wax-up into composite restorations without the need for tooth preparation. The injection molding technique has the advantage of replicating the excellent anatomy defined by a lab-made diagnostic wax-up whereby it would be used for the fabrication of direct restorations, so excellent anatomy results, verifies aesthetics, phonetics, and occlusion, avoids misunderstandings, as it is easy to implement and repair.

ELIGIBILITY:
Inclusion Criteria:

* Sound and vital upper anterior teeth.
* Spacing in the maxillary anterior teeth area ranging from .5mm to 2mm.
* Minor misalignment, correction of peg laterals.

Exclusion Criteria:

* Non-vital, fractured, or cracked teeth.
* Teeth with caries or in need of replacement of existing restorations.
* Rampant caries, atypical extrinsic staining of teeth.
* Heavy occlusion and occlusal contacts or history of bruxism.
* Severe periodontal affection.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Esthetic anatomical form at 6,12,18& 24 months. | T1: Baseline. T2: 6 months. T3: 12 months. T4: 18 months. T5: 24 months.
  FDI criteria. Possible scores range from 1 (Excellent) to 5 (Immediate replacement necessary).

SECONDARY OUTCOMES:
Change from baseline in Color match and translucency at 6,12,18& 24 months. | T1: Baseline. T2: 6 months. T3: 12 months. T4: 18 months. T5: 24 months.
  FDI criteria. Possible scores range from 1 (Excellent) to 5 (Immediate replacement necessary).
Change from baseline in Surface and marginal staining at 6,12,18& 24 months. | T1: Baseline. T2: 6 months. T3: 12 months. T4: 18 months. T5: 24 months.
  FDI criteria. Possible scores range from 1 (Excellent) to 5 (Immediate replacement necessary).
Change from baseline in Surface lustrous at 6,12,18& 24 months. | T1: Baseline. T2: 6 months. T3: 12 months. T4: 18 months. T5: 24 months.
  FDI criteria. Possible scores range from 1 (Excellent) to 5 (Immediate replacement necessary).